CLINICAL TRIAL: NCT04228848
Title: Examination of New Triple Hop Test Assessment Tool for Adults and Adolescents, Healthy and After Anterior Cruciate Ligament Injury
Brief Title: New Triple Hop Test Quality Assessment Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, Head of department of Physical therapy, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HU 1122
Record Dates: First submitted 2020-01-12; First posted 2020-01-14 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: 4 subgroups performing jump test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy adult (Active Comparator): Each participants will be asked to perform triple hop test on a straight line and to stand stable at the end of the jump. Two jumps will be performed on each leg, with 1 minute rest between them. The jumps will be recorded via video. Legs muscle strength will be assessed using hand held dynamometer
  Interventions: Other: new triple hop test
- ACL adult (Experimental): Each participants will be asked to perform triple hop test on a straight line and to stand stable at the end of the jump. Two jumps will be performed on each leg, with 1 minute rest between them. The jumps will be recorded via video. Legs muscle strength will be assessed using hand held dynamometer
  Interventions: Other: new triple hop test
- Healthy adolescent (Active Comparator): Each participants will be asked to perform triple hop test on a straight line and to stand stable at the end of the jump. Two jumps will be performed on each leg, with 1 minute rest between them. The jumps will be recorded via video. Legs muscle strength will be assessed using hand held dynamometer
  Interventions: Other: new triple hop test
- ACL adolescent (Experimental): Each participants will be asked to perform triple hop test on a straight line and to stand stable at the end of the jump. Two jumps will be performed on each leg, with 1 minute rest between them. The jumps will be recorded via video.Legs muscle strength will be assessed using hand held dynamometer
  Interventions: Other: new triple hop test

INTERVENTIONS:
Other: new triple hop test — New jumping assessment will be performed in all included study groups. This new assessment includes quality evaluation.

SUMMARY:
This study will develop a new jump assessment tool for the Triple Hop Test, and will test its reliability on adolescent and adult, healthy and post- anterior cruciate ligament (ACL) population.

Creating a new assessment test for a jump test that incorporates the known movement components that are important after an ACL injury can improve patient evaluation, decision for return to sport activity and injury prevention.

DETAILED DESCRIPTION:
Study population- Adults, women and men aged 20-45, boys and girls aged 12-15. uninjured population: non symptomatic subjects, without major injury in their history. Injured population: ACL injured subjects, 9-12 month after beginning of treatment/surgery.

Stages of study:

stage 1- The investigators will create a new high-quality literature-based assessment test for the triple hop test (NTHT). The test will have 10 sections, its score ranges from 0 to 14 points and a high score means poor performance.

Stage 2- Performing reliability tests between and within the testers for NTHT. The tests will be done with the help of video photography of NTHT.

Stage 3- Performing NTHT and THT tests on healthy adult and adolescent subjects and on ACL adult and adolescent subjects, assessing the NTHT by watching video performance.

ELIGIBILITY:
Inclusion Criteria uninjured population:

* non symptomatic subjects
* without major injury in their history.

Inclusion Criteria injured population:

* ACL injured subjects
* 9-12 month after beginning of treatment/surgery.

Exclusion Criteria uninjured population:

* acute pain
* knee instability symptoms
* history of lower leg injury
* unable to jump on one leg
* knee ligament injury.

Exclusion Criteria Injured population:

* late in rehabilitation program
* unable to jump or run
* instability symptoms.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
New triple hop test score | baseline
  the score ranges between 0-14. lower score represent better jumping quality.
triple hop test | baseline
  measurement of jumping distance(in cm) and symmetry between legs
muscle strength | baseline
  muscle strength in Newton, assessed by an hand held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
following study completion, a paper will be submitted to international professional journal
Supporting Information: Study Protocol, SAP
Time Frame: 6 months following end of study

REFERENCES:
- [Result] Graziano J, Chiaia T, de Mille P, Nawabi DH, Green DW, Cordasco FA. Return to Sport for Skeletally Immature Athletes After ACL Reconstruction: Preventing a Second Injury Using a Quality of Movement Assessment and Quantitative Measures to Address Modifiable Risk Factors. Orthop J Sports Med. 2017 Apr 20;5(4):2325967117700599. doi: 10.1177/2325967117700599. eCollection 2017 Apr. PMID 28451617
- [Result] Dekker TJ, Godin JA, Dale KM, Garrett WE, Taylor DC, Riboh JC. Return to Sport After Pediatric Anterior Cruciate Ligament Reconstruction and Its Effect on Subsequent Anterior Cruciate Ligament Injury. J Bone Joint Surg Am. 2017 Jun 7;99(11):897-904. doi: 10.2106/JBJS.16.00758. PMID 28590374